CLINICAL TRIAL: NCT00450437
Title: A Phase 3, Multi-center Study to Evaluate Lot to Lot Consistency, Safety and Immune Response of Novartis Meningococcal ACWY Conjugate Vaccine In US Adolescents and Adults and Compare to the Safety and Immune Response to a Licensed Conjugate Meningococcal ACWY Vaccine
Brief Title: A Study to Evaluate Safety and Immune Response of Novartis Meningococcal ACWY Conjugate Vaccine In US Adolescents and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V59P13
Record Dates: First submitted 2007-03-21; First posted 2007-03-22 (Estimated); Results first posted 2010-09-24 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Meningococcal Infections; Meningococcal Meningitis
Keywords: Meningococcal; meningitis; vaccine; adolescents; adults
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal; Meningitis | interventions — MenACWY-CRM vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Licensed Meningococcal Vaccine (Active Comparator): Licensed meningococcal ACWY polysaccharide-protein conjugate vaccine
  Interventions: Biological: Meningococcal ACWY Conjugate vaccine
- Novartis MenACWY Conjugate Vaccine (Experimental): Novartis meningococcal ACWY conjugate Vaccine
  Interventions: Biological: MenACWY CRM

INTERVENTIONS:
Biological: MenACWY CRM — One dose of the Novartis meningococcal ACWY conjugate vaccine was administered intramuscularly.
  Arms: Novartis MenACWY Conjugate Vaccine
Biological: Meningococcal ACWY Conjugate vaccine — One dose of the licensed meningococcal ACWY polysaccharide-protein conjugate vaccine was administered intramuscularly.
  Arms: Licensed Meningococcal Vaccine

SUMMARY:
This study will evaluate the lot to lot consistency, safety and immune response of the Novartis Meningococcal ACWY conjugate vaccine in healthy US adolescents and adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects who are 11-55 years of age inclusive and who have given appropriate written assent and/or consent

Exclusion Criteria:

* Subjects with a previous or suspected disease caused by N. meningitidis
* previous immunization with a meningococcal vaccine or vaccine containing meningococcal antigen(s)
* previous or suspected disease caused by N. meningitidis
* Any serious acute, chronic or progressive disease
* Pregnant or breastfeeding

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3539 (Actual)
Dates: Start 2007-03; Primary Completion 2007-08 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Director — Novartis
Locations (40):
- United States (40):
  - Birmingham, Alabama
  - Tuscaloosa, Alabama
  - Fremont, California
  - Fresno, California
  - Hayward, California
  - Oakland, California
  - Roseville, California
  - Sacramento, California
  - San Jose, California
  - Denver, Colorado
  - Atlanta, Georgia
  - Marietta, Georgia
  - Woodstock, Georgia
  - Chicago, Illinois
  - Bardstown, Kentucky
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Frederick, Maryland
  - Boston, Massachusetts
  - Fall River, Massachusetts
  - Lebanon, New Hampshire
  - Akron, Ohio
  - Cincinnati, Ohio
  - South Euclid, Ohio
  - Carnegie, Pennsylvania
  - Erie, Pennsylvania
  - Greenville, Pennsylvania
  - Grove City, Pennsylvania
  - Harleyville, Pennsylvania
  - Jefferson Borough, Pennsylvania
  - Latrobe, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Uniontown, Pennsylvania
  - Upper Saint Clair, Pennsylvania
  - Washington, Pennsylvania
  - Wexford, Pennsylvania
  - Galveston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington

REFERENCES:
- [Result] Jackson LA, Baxter R, Reisinger K, Karsten A, Shah J, Bedell L, Dull PM; V59P13 Study Group. Phase III comparison of an investigational quadrivalent meningococcal conjugate vaccine with the licensed meningococcal ACWY conjugate vaccine in adolescents. Clin Infect Dis. 2009 Jul 1;49(1):e1-10. doi: 10.1086/599117. PMID 19476428
- [Result] Reisinger KS, Baxter R, Block SL, Shah J, Bedell L, Dull PM. Quadrivalent meningococcal vaccination of adults: phase III comparison of an investigational conjugate vaccine, MenACWY-CRM, with the licensed vaccine, Menactra. Clin Vaccine Immunol. 2009 Dec;16(12):1810-5. doi: 10.1128/CVI.00207-09. Epub 2009 Oct 7. PMID 19812260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 44 centers in the US.
Pre-assignment Details: All subjects enrolled were included in the trial. All enrolled subjects were randomized at a 1:1:1:1 ratio to receive one of the four vaccine groups.
Groups:
- Novartis MenACWY Vaccine (11 to 18 Years); Novartis MenACWY Vaccine (19 to 55 Years): One dose of the Novartis meningococcal ACWY conjugate vaccine (obtained by extemporaneous mixing of components before injection) was administered intramuscularly.
- Licensed Meningococcal Vaccine (11 to 18 Years); Licensed Meningococcal Vaccine (19 to 55 Years): One dose of the licensed meningococcal ACWY polysaccharide-protein conjugate vaccine (supplied as a single 0.5 mL injection) was administered intramuscularly.
Period: Overall Study
Arm/Group | Novartis MenACWY Vaccine (11 to 18 Years) | Licensed Meningococcal Vaccine (11 to 18 Years) | Novartis MenACWY Vaccine (19 to 55 Years) | Licensed Meningococcal Vaccine (19 to 55 Years)
Started | 1640 | 540 | 1023 | 336
Completed | 1594 | 524 | 999 | 325
Not Completed | 46 | 16 | 24 | 11
Not completed — Withdrawal by Subject | 10 | 2 | 0 | 1
Not completed — Lost to Follow-up | 31 | 12 | 19 | 9
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Inappropriate enrollment | 4 | 1 | 3 | 0
Not completed — Administrative reason | 0 | 0 | 1 | 0
Not completed — Unable to Classify | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Novartis MenACWY Vaccine: One dose of the Novartis meningococcal ACWY (three lots combined) conjugate vaccine was administered intramuscularly.
- Licensed Meningococcal Vaccine: One dose of the licensed meningococcal ACWY polysaccharide-protein conjugate vaccine was administered intramuscularly.
- Total: Total of all reporting groups
Arm/Group | Novartis MenACWY Vaccine | Licensed Meningococcal Vaccine | Total
Number analyzed (Participants) | 2663 | 876 | 3539
Age, Continuous [Mean (Standard Deviation); unit: years]
  11 to 18 years | 14.2 (2.2) | 14.1 (2.2) | 14.2 (14.1)
  19 to 55 years | 39.0 (9.6) | 38.7 (9.9) | 39 (38.7)
Sex/Gender, Customized [Number; unit: participants]
  Female (11 to 18 years) | 769 | 251 | 1020
  Male (11 to 18 years) | 871 | 289 | 1160
  Female (19 to 55 years) | 774 | 252 | 1026
  Male (19 to 55 years) | 249 | 84 | 333
Race/Ethnicity, Customized [Number; unit: participants]
  Asian (11 to 18 years) | 45 | 17 | 62
  Black (11 to 18 years) | 138 | 45 | 183
  Caucasian (11 to 18 years) | 1280 | 423 | 1703
  Hispanic (11 to 18 years) | 126 | 34 | 160
  Other (11 to 18 years) | 51 | 21 | 72
  Asian (19 to 55 years) | 37 | 8 | 45
  Black (19 to 55 years) | 85 | 34 | 119
  Caucasian (19 to 55 years) | 828 | 261 | 1089
  Hispanic (19 to 55 years) | 60 | 29 | 89
  Other (19 to 55 years) | 13 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Lot to Lot Consistency of MenACWY as Measured by hSBA GMT Vaccine Group Ratios, Ages 11 to 18 Years
Description: The consistency of immune response for the three lots of Meningococcal ACWY (MenACWY), as measured by human serum bactericidal activity (hSBA) geometric mean titer (GMT) response using human complement (hSBA GMTs) directed against N. meningitidis serogroups A, C, W, and Y (healthy subjects 11 to 18 years of age)
Time Frame: 28 days after vaccination
Population: The analysis was performed on the Per Protocol (PP) Population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Novartis MenACWY Lot 1: One dose of the Novartis meningococcal ACWY conjugate Lot 1 vaccine was administered intramuscularly.
- Novartis MenACWY Lot 2: One dose of the Novartis meningococcal ACWY Lot 2 vaccine was administered intramuscularly.
- Novartis MenACWY Lot 3: One dose of the Novartis meningococcal ACWY Lot 3 vaccine was administered intramuscularly.
Arm/Group | Novartis MenACWY Lot 1 | Novartis MenACWY Lot 2 | Novartis MenACWY Lot 3
Number analyzed (Participants) | 359 | 357 | 359
Titers
  Serogroup A | 29 [23 to 38] | 33 [25 to 42] | 31 [24 to 40]
  Serogroup C (N=499, 493, 491) | 77 [58 to 102] | 58 [43 to 77] | 64 [48 to 86]
  Serogroup W (N=340, 341, 343) | 87 [70 to 108] | 111 [89 to 138] | 82 [66 to 102]
  Serogroup Y (N=345, 345, 346) | 48 [37 to 62] | 61 [47 to 79] | 53 [41 to 69]
Statistical Analysis 1: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain A at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 0.89, 95% CI 2-sided [0.68 to 1.16]
Statistical Analysis 2: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain A at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 0.95, 95% CI 2-sided [0.73 to 1.23]
Statistical Analysis 3: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain A at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 1.06, 95% CI 2-sided [0.81 to 1.38]
Statistical Analysis 4: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain C at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 1.2, 95% CI 2-sided [0.9 to 1.6]
Statistical Analysis 5: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain C at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 1.33, 95% CI 2-sided [1 to 1.77]
Statistical Analysis 6: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain C at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 0.9, 95% CI 2-sided [0.68 to 1.2]
Statistical Analysis 7: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain W at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 0.79, 95% CI 2-sided [0.63 to 0.97]
Statistical Analysis 8: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain W at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 1.06, 95% CI 2-sided [0.86 to 1.13]
Statistical Analysis 9: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain W at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval for all pairs of vaccine lots, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 1.35, 95% CI 2-sided [1.09 to 1.67]
Statistical Analysis 10: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain Y at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 0.79, 95% CI 2-sided [0.61 to 1.02]
Statistical Analysis 11: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain Y at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 0.91, 95% CI 2-sided [0.7 to 1.18]
Statistical Analysis 12: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; The study would be considered a success if the two-sided 95% confidence intervals (CIs) for the hSBA GMT ratios comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain Y at 1 month after vaccination was contained within the equivalence interval (0.5, 2.0); Test type: Non-Inferiority or Equivalence — The equivalence margin was (0.5, 2.0). If the two sided 95% CIs for the ratio of the hSBA GMT at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; hSBA GMT ratios = 1.16, 95% CI 2-sided [0.89 to 1.5]

2. Primary Outcome: Percentage of Seroresponders, Ages 11 to 18 Years
Description: Immunogenicity of a single injection of Meningococcal ACWY (3 lots pooled) to that of a licensed meningococcal ACWY conjugate vaccine, defined as the percentage of subjects with seroresponse directed against N meningitidis serogroups A, C, W, and Y (healthy adolescents 11 to 18 years of age).
  Seroresponse to MenACWY: For a subject with hSBA titer <1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer ≥ 1:8; for a subject with hSBA titer ≥ 1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 28 days after vaccination
Population: The analysis set was the per protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Novartis MenACWY Vaccine: One dose of the Novartis meningococcal ACWY (three lots combined)conjugate vaccine was administered intramuscularly.
- Licensed Meninogcoccal Vaccine: One vaccination of the licensed meningococcal ACWY polysaccharide-protein conjugate vaccine was administered intramuscularly.
Arm/Group | Novartis MenACWY Vaccine | Licensed Meninogcoccal Vaccine
Number analyzed (Participants) | 1075 | 359
Percentage of participants
  Serogroup A | 75 [72 to 77] | 66 [61 to 71]
  Serogroup C (N= 1483, 501) | 75 [73 to 77] | 73 [69 to 77]
  Serogroup W (N= 1024, 288) | 75 [72 to 77] | 63 [57 to 68]
  Serogroup Y (N= 1036, 294) | 68 [65 to 71] | 41 [35 to 47]
Statistical Analysis 1: Comparison: Novartis MenACWY Vaccine vs Licensed Meninogcoccal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenA; Test type: Non-Inferiority or Equivalence — Immunogenicity of the Investigational MenACWY vaccine would be considered non-inferior to that of the Licensed MenACWY vaccine if the lower limit of the two-sided CI for the between group difference (investigational vaccine minus licensed vaccine) in percentage of seroresponders one month after vaccination is > -10%; ANOVA; Vaccine group difference = 8, 95% CI 2-sided [3 to 14]
Statistical Analysis 2: Comparison: Novartis MenACWY Vaccine vs Licensed Meninogcoccal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; Vaccine group difference = 2, 95% CI 2-sided [-2 to 7]
Statistical Analysis 3: Comparison: Novartis MenACWY Vaccine vs Licensed Meninogcoccal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenW; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; Vaccine group difference = 12, 95% CI 2-sided [6 to 18]
Statistical Analysis 4: Comparison: Novartis MenACWY Vaccine vs Licensed Meninogcoccal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenY; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; Vaccine group difference = 27, 95% CI 2-sided [20 to 33]

3. Primary Outcome: Number of Participants With at Least One Severe Systemic Reaction, Ages 11 to 55 Years
Description: Safety of Novartis Meningococcal ACWY and of a licensed meningococcal ACWY conjugate vaccine as measured by the number of participants presenting at least one severe systemic reaction during the first 7 days (Days 1-7) following a single vaccination.
  Note: severe adverse events: unable to perform normal daily activity
Time Frame: 6 days after vaccination
Population: The analysis was performed on the safety set.
Measure: Number; unit: Participants
Groups:
- Novartis MenACWY Vaccine: One dose of the meningococcal ACWY (three lots combined)conjugate vaccine was administered intramuscularly.
Arm/Group | Novartis MenACWY Vaccine | Licensed Meningococcal Vaccine
Number analyzed (Participants) | 2649 | 875
Participants | 94 | 24
Statistical Analysis 1: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, safety; Test type: Non-Inferiority or Equivalence — MenACWY was considered noninferior to Menactra if the upper limit of the two-sided 95% CI of the difference in the percentage of subjects experiencing at least one severe systemic reaction [MenACWY minus Menactra] was less than 6%; ANOVA; Vaccine group difference = 1, 95% CI 2-sided [-1 to 2]

4. Secondary Outcome: Lot to Lot Consistency for the Percentage of Subjects With Seroresponse, Human Serum Bactericidal Activity (hSBA) Titer ≥ 1:8, and ≥ 1:4, Ages 11 to 18 Years
Description: The consistency of the immune response for three lots of Meningococcal ACWY, as measured by the percentage of subjects with seroresponse, hSBA titer ≥ 1:4 and ≥ 1:8, directed against N meningitidis serogroups A, C, W, and Y (healthy adolescents 11 to 18 years of age).
  Seroresponse to MenACWY: For a subject with hSBA titer <1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer ≥ 1:8; for a subject with hSBA titer ≥ 1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 28 days after vaccination
Population: The Analysis set was the per protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Novartis MenACWY Lot 1: One dose of the meningococcal ACWY Lot 1 conjugate vaccine was administered intramuscularly.
- Novartis MenACWY Lot 2: One dose of the meningococcal ACWY Lot 2 conjugate vaccine was administered intramuscularly.
- Novartis MenACWY Lot 3: One dose of the meningococcal ACWY Lot 3 conjugate vaccine was administered intramuscularly.
Arm/Group | Novartis MenACWY Lot 1 | Novartis MenACWY Lot 2 | Novartis MenACWY Lot 3
Number analyzed (Participants) | 359 | 357 | 359
Percentage of Participants
  Seroresponse in serogroup A | 71 [66 to 76] | 75 [70 to 79] | 77 [73 to 82]
  Seroresponse in serogroup C (N= 499, 493, 491) | 78 [74 to 82] | 73 [69 to 77] | 74 [70 to 78]
  Seroresponse in serogroup W (N= 340, 341, 343) | 74 [69 to 78] | 80 [75 to 84] | 70 [65 to 75]
  Seroresponse in serogroup Y (N= 345, 345, 346) | 66 [61 to 71] | 72 [67 to 77] | 65 [60 to 70]
  hSBA Titer ≥ 1:8 in serogroup A | 72 [67 to 77] | 76 [71 to 80] | 78 [74 to 82]
  hSBA Titer ≥ 1:8 in serogroup C (N= 499, 493, 491) | 86 [82 to 89] | 84 [81 to 87] | 83 [79 to 86]
  hSBA Titer ≥ 1:8 in serogroup W (N= 340, 341, 343) | 95 [92 to 97] | 97 [95 to 99] | 96 [93 to 98]
  hSBA Titer ≥ 1:8 in serogroup Y (N= 345, 345, 346) | 86 [82 to 89] | 89 [85 to 92] | 88 [85 to 92]
  hSBA Titer ≥ 1:4 in serogroup A | 76 [72 to 81] | 79 [74 to 83] | 81 [77 to 85]
  hSBA Titer ≥ 1:4 in serogroup C (N= 499, 493, 491) | 89 [86 to 91] | 88 [85 to 91] | 88 [85 to 91]
  hSBA Titer ≥ 1:4 in serogroup W (N= 340, 341, 343) | 95 [92 to 97] | 97 [95 to 99] | 97 [94 to 98]
  hSBA Titer ≥ 1:4 in serogroup Y (N= 345, 345, 346 | 89 [85 to 92] | 92 [89 to 95] | 93 [90 to 96]
Statistical Analysis 1: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain A were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -3, 95% CI 2-sided [-10 to 3]
Statistical Analysis 2: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain A were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -6, 95% CI 2-sided [-12 to 0]
Statistical Analysis 3: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain A were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -3, 95% CI 2-sided [-9 to 4]
Statistical Analysis 4: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain C were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 5, 95% CI 2-sided [0 to 10]
Statistical Analysis 5: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain C were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 4, 95% CI 2-sided [-1 to 10]
Statistical Analysis 6: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain C were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -1, 95% CI 2-sided [-6 to 5]
Statistical Analysis 7: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain W were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -6, 95% CI 2-sided [-13 to 0]
Statistical Analysis 8: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain W were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 4, 95% CI 2-sided [-3 to 11]
Statistical Analysis 9: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain W were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval for all pairs of vaccine lots, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 10, 95% CI 2-sided [4 to 17]
Statistical Analysis 10: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain Y were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -6, 95% CI 2-sided [-13 to 1]
Statistical Analysis 11: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain Y were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 1, 95% CI 2-sided [-6 to 8]
Statistical Analysis 12: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with seroresponse comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain Y were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for percentage of subjects with seroresponse at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 7, 95% CI 2-sided [0 to 14]
Statistical Analysis 13: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain A were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -3, 95% CI 2-sided [-10 to 3]
Statistical Analysis 14: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain A were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -6, 95% CI 2-sided [-12 to 0]
Statistical Analysis 15: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain A were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -3, 95% CI 2-sided [-9 to 4]
Statistical Analysis 16: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain C were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 2, 95% CI 2-sided [-3 to 6]
Statistical Analysis 17: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain C were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval for all pairs of vaccine lots, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 3, 95% CI 2-sided [-2 to 7]
Statistical Analysis 18: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain C were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 1, 95% CI 2-sided [-3 to 6]
Statistical Analysis 19: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain W were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval for all pairs of vaccine lots, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -2, 95% CI 2-sided [-5 to 1]
Statistical Analysis 20: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain W were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -1, 95% CI 2-sided [-4 to 2]
Statistical Analysis 21: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain W were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval for all pairs of vaccine lots, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 1, 95% CI 2-sided [-2 to 4]
Statistical Analysis 22: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain Y were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -3, 95% CI 2-sided [-8 to 2]
Statistical Analysis 23: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain Y were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -3, 95% CI 2-sided [-8 to 2]
Statistical Analysis 24: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:8 comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain Y were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:8 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 0, 95% CI 2-sided [-5 to 5]
Statistical Analysis 25: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain A were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -2, 95% CI 2-sided [-9 to 4]
Statistical Analysis 26: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain A were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -5, 95% CI 2-sided [-11 to 1]
Statistical Analysis 27: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain A were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain A with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -2, 95% CI 2-sided [-8 to 4]
Statistical Analysis 28: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain C were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 1, 95% CI 2-sided [-3 to 5]
Statistical Analysis 29: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain C were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 0, 95% CI 2-sided [-4 to 4]
Statistical Analysis 30: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain C were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain C with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 0, 95% CI 2-sided [-4 to 4]
Statistical Analysis 31: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain W were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval for all pairs of vaccine lots, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -2, 95% CI 2-sided [-5 to 1]
Statistical Analysis 32: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain W were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval for all pairs of vaccine lots, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -1, 95% CI 2-sided [-4 to 2]
Statistical Analysis 33: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain W were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval for all pairs of vaccine lots, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain W with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = 1, 95% CI 2-sided [-2 to 3]
Statistical Analysis 34: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 2; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 2 for Neisseria Meningitidis strain Y were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval for all pairs of vaccine lots, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 2 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -3, 95% CI 2-sided [-8 to 1]
Statistical Analysis 35: Comparison: Novartis MenACWY Lot 1 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 1 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain Y were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 1 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -4, 95% CI 2-sided [-9 to 0]
Statistical Analysis 36: Comparison: Novartis MenACWY Lot 2 vs Novartis MenACWY Lot 3; Lot-to-lot consistency would be concluded if the two-sided 95% confidence intervals (CIs) for the percentage of subjects with hSBA titer ≥1:4 comparing Investigational vaccine MenACWY Lot 2 to Investigational vaccine MenACWY Lot 3 for Neisseria Meningitidis strain Y were contained within the equivalence interval (-10%, 10%); Test type: Non-Inferiority or Equivalence — The equivalence margin was (-10%, 10%). If the two sided 95% CIs for the percentage of subjects with hSBA titer ≥1:4 at one month following vaccination was within this equivalence interval, Investigational vaccine MenACWY Lot 2 and Investigational vaccine MenACWY Lot 3 would be equivalent for Neisseria Meningitidis strain Y with respect to the immune response to the vaccine lot; ANOVA; Vaccine group difference = -1, 95% CI 2-sided [-5 to 3]

5. Secondary Outcome: Percentage of Subjects With Seroresponse, Human Serum Bactericidal Activity (hSBA) Titer ≥ 1:8, and hSBA Titer ≥ 1:4, Ages 11 to 55 Years
Description: Immunogenicity of a single injection of MenACWY (3 lots combined) to that of a licensed meningococcal ACWY conjugate vaccine, defined as the percentage of subjects with seroresponse directed against N meningitidis serogroups A, C, W, and Y (healthy subjects 11 to 55 years of age).
  Seroresponse to MenACWY: For a subject with hSBA titer <1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer ≥ 1:8; for a subject with hSBA titer ≥ 1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 28 days after vaccination
Population: The analyses set was performed on the per protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Novartis MenACWY Vaccine | Licensed Meningococcal Vaccine
Number analyzed (Participants) | 2038 | 680
Percentage of participants
  Seroresponse in serogroup A | 71 [69 to 73] | 67 [63 to 71]
  Seroresponse in serogroup C (N= 2444, 819) | 72 [70 to 74] | 67 [64 to 70]
  Seroresponse in serogroup W (N= 1508, 580) | 67 [64 to 69] | 52 [47 to 56]
  Seroresponse in serogroup Y (N= 1539, 600) | 64 [61 to 66] | 41 [37 to 45]
  hSBA≥1:8 in serogroup A | 72 [70 to 74] | 69 [65 to 72]
  hSBA≥1:8 in serogroup C (N= 2444, 819) | 83 [81 to 84] | 79 [76 to 82]
  hSBA≥1:8 in serogroup W (N= 1508, 580) | 95 [94 to 96] | 89 [86 to 91]
  hSBA≥1:8 in serogroup Y (N= 1539, 600) | 85 [83 to 87] | 70 [66 to 73]
  hSBA≥1:4 in serogroup A | 75 [74 to 77] | 73 [69 to 76]
  hSBA≥1:4 in serogroup C (N= 2444, 819) | 87 [86 to 88] | 85 [83 to 88]
  hSBA≥1:4 in serogroup W (N= 1508, 580) | 96 [95 to 97] | 91 [88 to 93]
  hSBA≥1:4 in serogroup Y (N= 1539, 600) | 90 [88 to 91] | 77 [74 to 81]
Statistical Analysis 1: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenA; Test type: Non-Inferiority or Equivalence — Immunogenicity of the Investigational MenACWY vaccine would be considered non-inferior to that of the Licensed MenACWY vaccine if the lower limit of the two-sided CI for percentage of subjects with seroresponse one month after vaccination is > -10%; ANOVA; Vaccine group difference = 4, 95% CI 2-sided [0 to 8]
Statistical Analysis 2: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; ANOVA; Vaccine group difference = 5, 95% CI 2-sided [1 to 9]
Statistical Analysis 3: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs.Licensed MenaCWY vaccine, MenW; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; ANOVA; Vaccine group difference = 15, 95% CI 2-sided [11 to 20]
Statistical Analysis 4: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenY; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; ANOVA; Vaccine group difference = 23, 95% CI 2-sided [19 to 28]
Statistical Analysis 5: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenA; Test type: Non-Inferiority or Equivalence — Immunogenicity of the Investigational MenACWY vaccine would be considered non-inferior to that of the Licensed MenACWY vaccine if the lower limit of the two-sided CI for percentage of subjects with hSBA ≥ 1:8 one month after vaccination is > -10%; ANOVA; Vaccine group difference = 4, 95% CI 2-sided [0 to 8]
Statistical Analysis 6: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 5]; ANOVA; Vaccine group difference = 3, 95% CI 2-sided [0 to 7]
Statistical Analysis 7: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenW; Test type: Non-Inferiority or Equivalence — Immunogenicity of the Investigational MenACWY vaccine would be considered non-inferior to that of the Licensed MenACWY vaccine if the lower limit of the two-sided CI for percentage of subjects with with hSBA ≥ 1:8 one month after vaccination is > -10%; ANOVA; Vaccine group difference = 6, 95% CI 2-sided [4 to 9]
Statistical Analysis 8: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenY; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 5]; ANOVA; Vaccine group difference = 15, 95% CI 2-sided [12 to 20]
Statistical Analysis 9: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenA; Test type: Non-Inferiority or Equivalence — Immunogenicity of the Investigational MenACWY vaccine would be considered non-inferior to that of the Licensed MenACWY vaccine if the lower limit of the two-sided CI for percentage of subjects with hSBA ≥ 1:4 one month after vaccination is > -10%; ANOVA; Vaccine group difference = 3, 95% CI 2-sided [-1 to 7]
Statistical Analysis 10: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 9]; ANOVA; Vaccine group difference = 1, 95% CI 2-sided [-1 to 4]
Statistical Analysis 11: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenW; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 9]; ANOVA; Vaccine group difference = 6, 95% CI 2-sided [3 to 8]
Statistical Analysis 12: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenY; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 9]; ANOVA; Vaccine group difference = 12, 95% CI 2-sided [9 to 16]

6. Secondary Outcome: Human Serum Bactericidal Activity (hSBA) Geometric Mean Titers, Ages 11 to 55 Years
Description: Immunogenicity of a single injection of MenACWY (3 lots combined) to that of a single injection of a licensed meningococcal ACWY conjugate vaccine, as measured by hSBA GMTs directed against N meningitidis serogroups A, C, W, and Y (healthy subjects 11 to 55 years of age).
Time Frame: 28 days after vaccination
Population: The analysis set was the per protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Novartis MenACWY Vaccine | Licensed Meningococcal Vaccine
Number analyzed (Participants) | 2038 | 680
Titers
  Titers in serogroup A | 29 [26 to 32] | 22 [19 to 26]
  Titers in serogroup C (N= 2444, 819) | 55 [49 to 62] | 39 [33 to 47]
  Titers in serogroup W (N= 1508, 580) | 100 [90 to 112] | 57 [49 to 66]
  Titers in serogroup Y (N= 1539 600) | 53 [47 to 60] | 21 [18 to 25]
Statistical Analysis 1: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Non-inferiority of Investigational MenACWY Vaccine vs. Licensed MenACWY vaccine, MenA. The study would be considered a success if the lower limit of the two-sided 95% CIs for the hSBA GMT ratios comparing Investigational MenACWY vaccine to Licensed MenACWY vaccine for Neisseria Meningitidis strain A at 1 month after vaccination was to be above 0.5; Test type: Non-Inferiority or Equivalence — The equivalence lower limit was 0.5. If the lower limit of two sided 95% CIs for the ratio of the hSBA GMT (GMT for investigational vaccine / GMT for licensed vaccine) at one month following vaccination was above this limit, Investigational MenACWY vaccine would be non-inferior to Licensed MenACWY vaccine for Neisseria Meningitidis strain A with respect to the immune response; ANOVA; hSBA GMT ratios = 1.32, 95% CI 2-sided [1.12 to 1.56]
Statistical Analysis 2: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Non-inferiority of Investigation MenACWY vaccine vs. Licensed MenACWY vaccine, MenC. The study would be considered a success if the lower limit of the two-sided 95% CIs for the hSBA GMT ratios comparing Investigational MenACWY vaccine to Licensed MenACWY vaccine for Neisseria Meningitidis strain C at 1 month after vaccination was to be above 0.5; Test type: Non-Inferiority or Equivalence — The equivalence lower limit was 0.5. If the lower limit of two sided 95% CIs for the ratio of the hSBA GMT (GMT for investigational vaccine / GMT for licensed vaccine) at one month following vaccination was above this limit, Investigational MenACWY vaccine would be non-inferior to Licensed MenACWY vaccine for Neisseria Meningitidis strain C with respect to the immune response; ANOVA; hSBA GMT ratios = 1.4, 95% CI 2-sided [1.17 to 1.67]
Statistical Analysis 3: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Non-inferiority of Investigational MenACWY vaccine vs. Licensed MenACWY vaccine, MenW. The study would be considered a success if the lower limit of the two-sided 95% CIs for the hSBA GMT ratios comparing Investigational MenACWY vaccine to Licensed MenACWY vaccine for Neisseria Meningitidis strain W at 1 month after vaccination was to be above 0.5; Test type: Non-Inferiority or Equivalence — The equivalence lower limit was 0.5. If the lower limit of two sided 95% CIs for the ratio of the hSBA GMT (GMT for investigational vaccine / GMT for licensed vaccine) at one month following vaccination was above this limit, Investigational MenACWY vaccine would be non-inferior to Licensed MenACWY vaccine for Neisseria Meningitidis strain W with respect to the immune response; ANOVA; hSBA GMT ratios = 1.76, 95% CI 2-sided [1.51 to 2.05]
Statistical Analysis 4: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Non-inferiority of Investigational MenACWY Vaccine vs. Licensed MenACWY vaccine, MenY. The study would be considered a success if the lower limit of the two-sided 95% CIs for the hSBA GMT ratios comparing Investigational MenACWY vaccine to Licensed MenACWY vaccine for Neisseria Meningitidis strain Y at 1 month after vaccination was to be above 0.5; Test type: Non-Inferiority or Equivalence — The equivalence lower limit was 0.5. If the lower limit of two sided 95% CIs for the ratio of the hSBA GMT (GMT for investigational vaccine / GMT for licensed vaccine) at one month following vaccination was above this limit, Investigational MenACWY vaccine would be non-inferior to Licensed MenACWY vaccine for Neisseria Meningitidis strain Y with respect to the immune response; ANOVA; hSBA GMT ratios = 2.49, 95% CI 2-sided [2.11 to 2.95]

7. Secondary Outcome: Number of Subjects With Local and Systemic Reactions, Ages 11 to 55 Years
Description: Safety profile following a single injection of MenACWY (3 lots combined) was to that following a single injection of a licensed meningococcal ACWY conjugate vaccine administered to healthy adolescents or adults (11 to 55 years of age).
Time Frame: Days 1 to 7
Population: The analysis was performed on the safety set.
Measure: Number; unit: Participants
Arm/Group | Novartis MenACWY Vaccine | Licensed Meningococcal Vaccine
Number analyzed (Participants) | 2649 | 875
Participants
  Pain | 1105 | 424
  Erythema | 414 | 126
  Induration | 324 | 88
  Chills | 168 | 50
  Nausea | 260 | 65
  Malaise | 279 | 99
  Myalgia | 452 | 149
  Arthralgia | 197 | 54
  Headache | 731 | 237
  Rash | 69 | 20
  Fever ≥38°C | 32 | 6
  Any Other Reaction | 555 | 183
  Analgesic/Antipyretic Medication Used | 533 | 178
  Stayed Home | 69 | 17

8. Primary Outcome: Percentage of Seroresponders, Ages 19 to 55 Years
Description: Immunogenicity of a single injection of Meningococcal ACWY (3 lots pooled) to that of a licensed meningococcal ACWY conjugate vaccine, defined as the percentage of subjects with seroreponse directed against N. meningitidis serogroups A, C, W, and Y (healthy subjects 19 to 55 years of Age).
  Seroresponse to MenACWY: For a subject with hSBA titer <1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer ≥ 1:8; for a subject with hSBA titer ≥ 1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 28 days after vaccination
Population: The analysis set was the per protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Novartis MenACWY Vaccine | Licensed Meningococcal Vaccine
Number analyzed (Participants) | 963 | 321
Percentage of participants
  Serogroup A | 67 [64 to 70] | 68 [63 to 73]
  Serogroup C (N=961, 318) | 67 [64 to 70] | 58 [53 to 64]
  Serogroup W (N= 484, 292) | 50 [46 to 55] | 41 [35 to 47]
  Serogroup Y (N= 503, 306) | 56 [51 to 60] | 40 [34 to 46]
Statistical Analysis 1: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenA; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; Vaccine group difference = -1, 95% CI 2-sided [-7 to 5]
Statistical Analysis 2: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine. MenC; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; Vaccine group difference = 9, 95% CI 2-sided [3 to 15]
Statistical Analysis 3: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenW; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; Vaccine group difference = 9, 95% CI 2-sided [2 to 17]
Statistical Analysis 4: Comparison: Novartis MenACWY Vaccine vs Licensed Meningococcal Vaccine; Vaccine group difference Investigational MenACWY vaccine vs. Licensed MenaCWY vaccine, MenY; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; Vaccine group difference = 16, 95% CI 2-sided [9 to 23]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from study day 1 to 180.
Description: A total of 3539 subjects were enrolled in the study; 3524 were vaccinated to receive MenACWY (2649 subjects) or Menactra (875). ). Overall, 15 subjects were not vaccinated and were excluded from the safety analysis.
Groups:
- Novartis MenACWY Vaccine: One dose of the Novartis meningococcal ACWY conjugate vaccine (three lots combined) was administered intramuscularly, 11 to 55 years of age.
- Licensed Meningococcal Vaccine: One dose of the licensed meningococcal ACWY polysaccharide-protein conjugate vaccine was administered intramuscularly, 11 to 55 years of age.
Arm/Group | Novartis MenACWY Vaccine | Licensed Meningococcal Vaccine
Serious Adverse Events (participants affected / at risk) | 23/2649 | 5/875
Other Adverse Events (participants affected / at risk) | 1613/2649 | 572/875
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novartis MenACWY Vaccine (N=2649) | Licensed Meningococcal Vaccine (N=875)
Vitello-Intestinal Duct Remnant (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis Viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns Second Degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dislocation of Sternum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epishysiolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonic Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Simple Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Depression Suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Circulatory Collapse (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Novartis MenACWY Vaccine (N=2649) | Licensed Meningococcal Vaccine (N=875)
Injection site pain (General disorders) | 1106 | 424
Injection site erythema (General disorders) | 414 | 126
Injection site induration (General disorders) | 324 | 88
Chills (General disorders) | 169 | 50
Nausea (Gastrointestinal disorders) | 265 | 66
Malaise (General disorders) | 280 | 100
Myalgia (Musculoskeletal and connective tissue disorders) | 453 | 150
Arthralgia (Musculoskeletal and connective tissue disorders) | 211 | 59
Headache (Nervous system disorders) | 740 | 240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No